CLINICAL TRIAL: NCT05412264
Title: Step Up for Health: A Pedometer-based Randomized Controlled Trial for Individuals at High Risk for Type 2 Diabetes
Brief Title: Step Up For Health Study: A Pedometer and Website Intervention in Those With Prediabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: REB Approval lapsed.
Sponsor: University of Alberta (Other)
Collaborators: Athabasca University (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00039828
Record Dates: First submitted 2015-01-21; First posted 2022-06-09 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-05

CONDITIONS: Prediabetes; Impaired Glucose Tolerance
Keywords: Prediabetes; Pedometer; Web-based
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Website intervention (Experimental): Website access: 12 Weekly emails, access to website with goal setting and recording steps
  Interventions: Behavioral: Website intervention
- Delayed access (No Intervention): Will not receive access to the program/website until they complete their 16 week assessments

INTERVENTIONS:
Behavioral: Website intervention — 12 week motivational emails, recording pedometer steps and waist circumference
  Arms: Website intervention

SUMMARY:
This study will examine whether a physical activity program, specifically increasing walking steps, offered over the internet is able to increase physical activity in adults with prediabetes. The study will take place over 12 weeks. The investigators want to see if people who receive the intervention increase their physical activity more than people who do not receive the intervention. The physical activity program will include using a pedometer to track daily step counts online, set weekly goals, and receive motivational messages delivered weekly using email. The investigators are also going to collect data on waist circumference, body weight and quality of life at baseline, 12 weeks and 16 weeks after the intervention has completed to see if these change over the course of the study. The investigators will be recruiting 200 adults who have attended the Edmonton, Alberta prediabetes education class offered by Alberta Health Services, Nutrition Services and report they have prediabetes. If able to successfully increase physical activity, this study will identify a web and home-based intervention that can be offered to individuals who participate in lifestyle programs delivered in primary care settings (e.g., Edmonton prediabetes program) in both rural and urban locations.

DETAILED DESCRIPTION:
Relevance to diabetes: Without intervention, most people at high-risk of diabetes (e.g., with prediabetes) will eventually develop type 2 diabetes over time. Moderate physical activity of 150 minutes per week has been demonstrated to improve glucose tolerance and decrease type 2 diabetes risk. Research is needed to determine the effectiveness and acceptability of web-based methods of increasing physical activity, specifically walking, in these high risk populations.

Brief background of the issue: Studies completed in adults with prediabetes have demonstrated lower physical activity levels than the general population; however, adults with prediabetes have reported they are interested in a physical activity program that is focused on individuals with prediabetes.

Objective: To determine if a theoretically-based physical activity internet website with pedometer step and physical activity monitoring is able to increase physical activity behavior among adults at high risk of type 2 diabetes.

Hypothesis: Individuals at high risk of type 2 diabetes randomized to the intervention group will increase their pedometer steps and physical activity over a 12-week intervention compared to individuals in the control group.

Methods: Four hundred adults at high risk of type 2 diabetes will be recruited from the Edmonton and Calgary prediabetes education classes by Registered Dietitians (RD) teaching the class. The RD will discuss the study and interested participants will receive a pedometer, waist circumference tape and study information letter at the class. In the study information letter they will be directed to a website where they can agree to participate in the study after completing a brief questionnaire to determine study eligibility and a Physical activity readiness (e-ParMedX) form to determine physical activity safety. After completing these documents, if they are eligible to participate they will complete an online baseline questionnaire, a 3-day pedometer step test and a waist circumference measurement. All measurements and personal information will be recorded on the secure website. These measurements will be repeated at 12 weeks and 16 weeks post intervention. Upon completion of the baseline measures, they will be randomized by the website program into either the control or intervention group. The intervention group will receive a theoretically-based 12-week intervention program via the website designed to increase their physical activity and steps. The website content is based on the theory of planned behaviour and tailored to people at high-risk of type 2 diabetes. Participants will receive weekly information that is temporally sequenced on the website for each of the 12 weeks, set weekly goals and record their daily steps on the website. After the control group has completed their six-month assessment they will also be able to access the 12 week intervention.

Application to Practice: If able to successfully increase physical activity, this trial will identify a theoretically-based web and home-based intervention that can be offered to individuals who participate in lifestyle programs delivered in primary care settings (e.g., Edmonton prediabetes program) in both rural and urban locations. Research is needed to determine the effectiveness and acceptability of web-based methods of increasing physical activity, specifically walking, in these high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* You are over 18 years of age.
* Have been told you have prediabetes by a health professional.
* You are free from any medical problems that make it hard to be active. For example, congestive heart failure, a recent knee or hip replacement, or you need to use a cane or walker to help you walk.
* Live in Alberta.
* Are interested in finding ways to become more physically active.
* Are interested in wearing a pedometer and tracking your daily steps.

Exclusion Criteria:

* You have been told you have type 2 diabetes.
* You do not confirm on the website that it is safe for you to increase your walking or other physical activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10-05 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Increased pedometer steps | 12 weeks
  Measured as a 3-day step test
Increased pedometer steps | 16 weeks
  Measured as a 3-day step test

SECONDARY OUTCOMES:
Waist circumference | 12 weeks
  Measured
Waist circumference | 16 weeks
  Measured

OTHER OUTCOMES:
Questionnaire | 12 weeks
  Measuring changes in attitude, social norms and perceived behavioral control
Questionnaire | 16 weeks
  Measuring changes in attitude, social norms and perceived behavioral control

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Vallance, PhD, Principal Investigator — Athabasca University; Lorian Taylor, PhD, Principal Investigator — Alberta Health services
Locations (1):
- Alberta Health Services, Nutrition Services, Edmonton, Alberta, Canada